CLINICAL TRIAL: NCT05162274
Title: An Open-label, Randomized, Fasted, Single-dose, Oral Administration, 2-sequence, 2-period Crossover Study to Assess Bioequivalence of Lazertinib Between Two Formulations in Healthy Adult Volunteers
Brief Title: Clinical Trial to Assess Bioequivalence of Lazertinib Between Two Formulations in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH25448-102
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2022-02

CONDITIONS: Healthy Adult Volunteers
Keywords: YH25448; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Participants first received lazertinib(G001) 240mg tablet morning in a fasting state for 1 day. After a washout period of 14~21days, they then received lazertinib(G002) 240mg in a fasting state morning for 1 day.
  Interventions: Drug: Lazertinib(G001); Drug: Lazertinib(G002)
- Group 2 (Experimental): Participants first received lazertinib(G002) 240mg tablet morning in a fasting state for 1 day. After a washout period of 14~21days, they then received lazertinib(G001) 240mg in a fasting state morning for 1 day.
  Interventions: Drug: Lazertinib(G001); Drug: Lazertinib(G002)

INTERVENTIONS:
Drug: Lazertinib(G001) — Current formulation
Drug: Lazertinib(G002) — New formulation

SUMMARY:
This Clinical Trial is an open, randomized, fasted, single-dose, oral administration 2-sequence, 2-period crossover study to assess bioequivalence of lazertinib between two formulations in healthy adult volunteers. The subjects administer 240mg of lazertinib of different formulations on the fasted status on each period and have a wash-out period for 14-21 days between the first and second period.

DETAILED DESCRIPTION:
This clinical trial will be conducted in healthy male volunteers at Seoul National University Hospital (SNUH) Clinical Trial Center.

It is expected to take approximately 32 days from the first dosing of Investigational Product until the final follow-up visit. Subjects will be hospitalized twice for 4 nights and 5 days with 7-14 days of wash-out period, and one visit will be needed for safety evaluation between 14-17 days from the last dosing of the Investigational Product.

ELIGIBILITY:
Inclusion Criteria:

* Male, over 19 years of age
* Male participants must agree to use an adequate contraception method from the first to the third month after the last dose.
* Participants must have a body mass index (BMI) between 18.5 and 30.0 kg/m2, inclusive(BMI = weight/height2), and body weight not less than 50 kg.
* Subjects without congenital or chronic diseases within the last 3 years and without pathologic symptoms as determined by medical diagnosis.
* Participants must be healthy on the basis of clinical laboratory tests performed at screening.
* Informed of the investigational nature of this study and voluntarily agree to participate in this study.

Exclusion Criteria:

* Clinically significant medical or psychiatric illness.
* Hypotension (SBP ≤ 90 mmHg or DBP ≤ 50 mmHg) or hypertension (SBP ≥ 150 mmHg or DBP ≥ 100 mmHg).
* A marked baseline prolongation of QTc.
* Within 14 days prior to the first administration of investigational product, use of prescription drugs or herbal medication, or within 7 days use of any over-the-counter medications
* Participants who are planning COVID-19 vaccine within 14 days before the first intake of study drug and to the end of the trials.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
AUClast of YH25448 | 0 - 168 hours
  Area under the plasma concentration-time curve from zero to the time of the last quantitative concentration (AUC) of YH25448
Cmax of YH25448 | 0 - 168 hours
  Area under the plasma concentration-time curve from zero to the time of Maximum plasma concentration (Cmax) of YH25448

SECONDARY OUTCOMES:
AUC0-72h of YH25448 | 0 - 72 hours
  Area under the plasma concentration-time curve from zero to the time of the last quantitative concentration (AUC) of YH25448
AUCinf of YH25448 | 0 - 168 hours
  Area under the plasma concentration time curve from zero to infinity (AUC) of YH25448
Tmax of YH25448 | 0 - 168 hours
  Time to reach Cmax of YH25448
t1/2 of YH25448 | 0 - 168 hours
  Terminal half life (t1/2) of YH25448
λz of YH25448 | 0 - 168 hours
  Terminal rate constant of YH25448
CL/F of YH25448 | 0 - 168 hours
  The apparent plasma clearance (CL/F) of YH25448
Vd/F of YH25448 | 0 - 168 hours
  Apparent Volume of distribution of YH25448

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development and Medical Department, Study Director — Yuhan Corporation
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No